CLINICAL TRIAL: NCT05743140
Title: A Clinical Study of Fundus Optical Coherence Tomography Angiography for the Identification of Coronary Microvascular Diseases
Brief Title: A Clinical Study of Fundus OCTA for the Identification of CMD
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, ZHENG Bo, associate professor, Peking University First Hospital
Other Study IDs: ZHENG Bo
Record Dates: First submitted 2023-02-07; First posted 2023-02-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Coronary Microvascular Disease
Keywords: coronary microvascular disease; CaIMR; OCT; OCTA; Fundus microcirculation
MeSH Terms: conditions — Microvascular Angina

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CMD group, Non-CMD group: CMD group: participants whose CaIMR shows ≥25U. Non-CMD group: participants whose CaIMR less than 25U.
  Interventions: Diagnostic Test: CaIMR

INTERVENTIONS:
Diagnostic Test: CaIMR — Investigators diagnose CMD with CaIMR. Investigators use OCT and OCTA to analyze the fundus microcirculation quantitatively.
  Other Names: OCT; OCTA

SUMMARY:
Coronary microvascular dysfunction (CMD) carries an increased risk of adverse cardiovascular clinical outcomes. The association between fundus microcirculation changes and coronary microcirculation is not well understood. Optical coherence tomography (OCT) and optical coherence tomography angiography (OCTA) is a new type of optical diagnostic imaging technology for non-invasive detection, which can perform multi-dimensional quantitative assessment of fundus microcirculation. In this study, investigators intend to use the coronary angiography-derived index of microvascular resistance (caIMR) to screen patients with CMD, explore the relationship between relevant parameters based on OCT and OCTA measurements and caIMR, and evaluate the feasibility and clinical value of non-invasive identification of CMD through fundus OCT and OCTA.

DETAILED DESCRIPTION:
Coronary microvascular dysfunction (CMD) is defined as the clinical syndrome of angina and electrocardiographic ischemic changes in the absence of obstructive coronary artery disease. CMD carries an increased risk of adverse cardiovascular clinical outcomes. Assessment of CMD is performed with different diagnostic modalities, including nuclear myocardial scintigraphy, cardiac magnetic resonance, doppler echocardiography, and coronary microcirculation resistance index techniques. However, current examination techniques have limitations such as radiation risk, high cost, and time-consuming, so they cannot be widely screened in the population. Previous studies have shown that fundus vascular changes were strongly associated with cardiovascular events, but the correlation between fundus microcirculation changes and coronary microcirculation is not well understood. Optical coherence tomography (OCT) and optical coherence tomography angiography (OCTA) is a new type of optical diagnostic imaging technology for non-invasive detection, which use infrared light projection onto fundus tissue to achieve real-time tomographic section imaging, which can perform multi-dimensional quantitative assessment of fundus microcirculation. In this study, investigators intend to use the coronary angiography-derived index of microvascular resistance (caIMR) to screen patients with CMD, explore the relationship between relevant parameters based on OCT and OCTA measurements and caIMR, and evaluate the feasibility and clinical value of non-invasive identification of CMD through fundus OCT and OCTA.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent coronary angiography in the Department of Cardiology, Peking University First Hospital;
2. Complete baseline clinical information;
3. Subject who have coronary angiography results, which shows coronary stenosis < 50%;
4. Older than 18 years;
5. Subjects who have signed informed consent.

Exclusion Criteria:

1. Present serious fundus disease
2. Severe cataract and other ophthalmic diseases, which affect imaging quality;
3. Target coronary vessels provide collateral circulation for chronic complete occlusive lesions;
4. The target coronary angiography agent is poorly filled, overlapped, or severely distorted, and cannot fully expose the location of the lesion;
5. Coronary angiography images are of poor quality and cannot be identified;
6. Active bleeding state;
7. Severe renal insufficiency, contrast agent allergy, and unable to perform coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Department of Cardiology, Peking University First Hospital
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of fundus OCT and OCTA examinations for coronary microvascular disease | 2023.3-2024.5
  Investigators intend to use these indicators to assess the diagnostic accuracy of fundus OCT and OCTA for CMD: area under the receiver operating characteristic curve (AUROC), sensitivity, specificity, positive likelihood ratio, and negative likelihood ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Zheng, Dr, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking university first hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No